CLINICAL TRIAL: NCT02213523
Title: Proof of Concept Study to Evaluate the Effect of Oxidative Stress Response of Plant Concentrate Blends in Healthy Men
Brief Title: ABG Oxidative Stress Study Protocol-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABG AOX-1
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: antioxidant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Plant concentrate A (Experimental): Plant concentrate A containing Rosemary:Quercetin:Turmeric 5:3:1 Low dose (300 mg) to high dose (600 mg)
  Interventions: Dietary Supplement: Plant concentrate A
- Plant concentrate B (Experimental): Plant concentrate B containing Holy Basil: Wasabi: Broccoli 5:5:1 Low dose (300 mg) to high dose (600 mg)
  Interventions: Dietary Supplement: Plant concentrate B
- Plant concentrate C (Experimental): Plant concentrate C containing Holy Basil:Rosemary:Broccoli seed:Turmeric 2:2:1:1 Low dose (300 mg) to High dose (600 mg)
  Interventions: Dietary Supplement: Plant concentrate C
- Plant concentrate D (Experimental): Plant concentrate D containing Rosemary:Licorice:Turmeric 1:1:1 Low dose (300 mg) to High dose (600 mg)
  Interventions: Dietary Supplement: Plant concentrate D

INTERVENTIONS:
Dietary Supplement: Plant concentrate A — Screening for the optimal dosage by starting with with a low dose of 300 mg for one week then switch to 600 mg for one week.
  Arms: Plant concentrate A
Dietary Supplement: Plant concentrate B — Screening for the optimal dosage by starting with with a low dose of 300 mg for one week then switch to 600 mg for one week.
  Arms: Plant concentrate B
Dietary Supplement: Plant concentrate C — Screening for the optimal dosage by starting with with a low dose of 300 mg for one week then switch to 600 mg for one week.
  Arms: Plant concentrate C
Dietary Supplement: Plant concentrate D — Screening for the optimal dosage by starting with with a low dose of 300 mg for one week then switch to 600 mg for one week.
  Arms: Plant concentrate D

SUMMARY:
This is a proof of concept study that evaluates the response to oxidative stress in healthy men after taking plant concentrates.

DETAILED DESCRIPTION:
Sustained oxidative stress may cause hypertension, insulin resistance, metabolic syndrome, cardiovascular disease and other chronic conditions. Diets rich in natural antioxidants is associated with protective effects on the investigators health. The strategy to prevent chronic disease development and in making up the nutritional gap in the investigators diet has shifted from vitamins and minerals supplementation to whole foods and whole food products.

The objectives is to evaluate the effect of oxidative stress response of plant concentrate blends. Also, we'll confirm that vitamins, minerals and plant concentrates will not influence the biomarker expression that were monitored in the oxidative stress biomarkers. Lastly, collecting additional information on whether blends of plant concentrate have other potential health benefits.

This study will test the dose-response of blends of plant concentrates. Healthy men (n=60) with low fruit and vegetable intake will participate in a 32 day or 46 days. Each treatment duration lasts 14 days. Microarray assay and real time-polymerase chain reaction will be performed.Genes associated with oxidative stress will me monitored. The outcome of this study will help us understand how to design and develop future antioxidant related products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men between 45-65 yr old with low fruit and vegetable intake
* Individual with low fruit and vegetable intake and consuming fewer than 12 items found on the Recommended Foods Check (RFC) (AppendixI) per week. (score <12 pts)
* Individuals with screening blood and urine laboratory values within 20% of normal range indicated in the lab report (Appendix IV)
* Individual should be judged to be in good general health on the basis of an interview and abbreviated physical exam.
* Individual understands the procedures and agrees to participate in the study.
* Individual is willing to maintain their exercise habits and dietary pattern throughout the duration of the trial.
* Individual is willing to consume a diet or drink devoid of high content of quercetin (e.g. apple and onions), rosemary, turmeric, Holy basil, wasabi, broccoli seeds, and licorice thought the duration of the trial.
* Individual is able and willing to provide written informed consent and confidentiality agreement.

Exclusion Criteria:

* Use of dietary supplements within one week of DAy 1. Supplements include any vitamins, minerals, and herbal products, including herbal drink.
* Presence of, or clinical significant history of, cancer, cardiovascular, endocrine, kidney, liver, lung, gastrointestinal, metabolic disorder, absorption disorder such as Celiae or Crohn's disease and/or any other chronic health condition such as diabetes identified from the finding of the interview.
* Presence of cardiovascular disease and hypertension with inconsistent medication regimen, unstable conditions, and without proper physician's supervision identified from the findings fo the interview.
* Individual who use medicines such as statins (e.g. simvastatin, fluvastatin), NSAIDS including aspirin, nitric oxide *eNOS) activators or inhibitors (e.g. selegiline, Viagra), and angiotensin II receptor blocker (e.g. Telmisartan (blood pressure)), and take any of these medications within 10 hours prior to the blood and urine sample collection.
* Individuals who eat spicy food (e.g. capsaicin from chili pepper) and drink coffee and tea including herbal teas within 10 hours prior to the blood and urine sample collection.
* Participation in another clinical trial within 30 days of enrollment into the study.
* History of current abuse of nicotine, drugs or alcohol, or intake >3 alcoholic beverages per day
* Have known allergy to the ingredients in the tested samples such as quercetin, rosemary, turmeric, Holy basil, wasabi, broccoli seeds, and licorice.
* Any condition that the principal Investigator believes amy put the subject under risk.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in urine 8-isoprostane | Day 1, 15
  Change in antioxidant biomarker from baseline to day 15

SECONDARY OUTCOMES:
Change in erythrocyte Superoxide Dismutase | 1, 15
  Change in antioxidant biomarker from baseline to day 15
Change in plasma malondialdehyde | Day 1, 15
  Change in antioxidant biomarker from baseline to day 15
Plasma hemoxygenase-1 | Day 1, 15
  Change in antioxidant biomarker from baseline to day 15
Erythrocyte glutathione peroxidase | Day 1, 15
  Change in antioxidant biomarker from baseline to day 15

CONTACTS AND LOCATIONS:
Overall Officials: Richard Keech, M.D., Principal Investigator — Southbay Pharma Research
Locations (2):
- United States (2):
  - Quality of Life, Buena Park, California
  - Southbay Pharma Research, Buena Park, California